CLINICAL TRIAL: NCT04797000
Title: A Randomized, Double-blind, Placebo-controlled, Japan Local Phase II Clinical Study Comparing Eltrombopag Monotherapy Versus Placebo in Adult Lower-risk Myelodysplastic Syndromes (MDS) Patients With Platelet Transfusion Dependence
Brief Title: Study of Efficacy and Safety of Eltrombopag in Lower-risk MDS Patients With Platelet Transfusion Dependence
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CETB115L11201
Record Dates: First submitted 2021-03-04; First posted 2021-03-15 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: Phase II; eltrombopag; ETB115; lower-risk MDS patients with platelet transfusion dependence; TPO-RA; placebo; myelodysplastic syndromes (MDS); platelet transfusion dependence
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, site staffs and site monitors will remain blinded to the identity of the treatment from the time of randomization until database lock for final analysis, and the clinical study team members and anyone involved in the Japan registration activities will be blinded until database lock for the primary analysis. Randomization data are kept strictly confidential until the time of unblinding and will not be accessible by anyone else involved in the study with the following exceptions: DMC members and who will perform data analysis for DMC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eltrombopag Arm (Experimental): Participants randomized to a 1: 1 ratio will take eltrombopag.
  Interventions: Drug: Eltrombopag
- Placebo Arm (Placebo Comparator): Participants randomized to a 1: 1 ratio will take Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag comes in 12.5 mg & 25 mg tablets and is taken orally once per day (QD)
  Other Names: ETB115
  Arms: Eltrombopag Arm
Drug: Placebo — Placebo comes in 12.5 mg & 25 mg tablets and is taken orally once per day (QD)
  Arms: Placebo Arm

SUMMARY:
This study is designed to evaluate the efficacy and safety of eltrombopag monotherapy in Japanese adult patients with platelet transfusion-dependent lower-risk Myelodysplastic syndromes (LR-MDS).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, Japanese local phase II study to evaluate the efficacy and safety of eltrombopag monotherapy in Japanese adult patients with platelet transfusion-dependent lower-risk MDS (IPSS-R very low, low, intermediate risk with bone marrow blast count < 5% and cytogenetic very good, good or intermediate risk). Platelet transfusion dependence at baseline is defined as receiving platelet transfusion regularly with a frequency of 2 or more times within 4 weeks prior to randomization. Platelet transfusion should be performed for a patient with platelet counts < 20 X 10^9/L, or with hemorrhagic symptoms and platelet counts < 30 X 10^9/L.

The primary objective is to demonstrate superiority of eltrombopag versus placebo in terms of the proportion of participants who achieve platelet transfusion independence at Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with MDS according to the WHO classification revised 4th edition by investigator assessment with one of the following prognostic risk categories, based on the International

Prognostic Scoring System (IPSS-R):

* very low (0-1.5)
* low (2-3)
* intermediate risks (3.5-4.5) All following criteria for prognostic variables per IPSS-R should be met.
* Bone marrow blast < 5% (per both investigator's assessment and central review)
* Cytogenetic very good, good or intermediate risk corresponding to IPSS-R

  * Platelet transfusion dependence
  * Refractory, intolerant to, or ineligible for MDS treatments
  * Eastern Cooperative Oncology Group (ECOG) Performance status (PS) 0 or 1

Exclusion Criteria:

* Patients with a history of prior administration of eltrombopag, romiplostim, or other TPO-RA
* Therapy-related MDS per WHO classification revised 4th edition
* MDS/myeloproliferative neoplasms including chronic myelomonocytic leukaemia per the WHO classification revised 4th edition
* MDS with excess blasts (EB) per WHO classification revised 4th edition
* Known history of IPSS-R high or very high risk MDS
* Currently receiving treatments for MDS (e.g., HMA, cyclosporine A (CsA) or lenalidomide). Supportive treatment with erythropoiesis-stimulating agents (ESAs) in anemic patients or granulocyte-colony stimulating factor (G-CSF) in patients with severe neutropenia and recurrent infections is allowed if at stable dosage for 3 months prior to screening and continued at the same dosing/schedule until the optimal dose of eltrombopag has been established.
* Patients scheduled for hematopoietic stem cell transplantation
* Bone marrow fibrosis that leads to an inability to aspirate adequate bone marrow sample
* Known thrombophilic risk factors (except in cases where potential benefits of participating in the study outweighed potential risks of thromboembolic events(TEE), as determined by the investigator)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2025-04-26 (Actual); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who achieve platelet transfusion independence at Week 24 | Week 24
  Platelet transfusion independence is defined as the absence of platelet transfusion for at least 8 weeks. Platelet count should be higher than the baseline count.

SECONDARY OUTCOMES:
Time to platelet transfusion independence | Year 1, Year 2
  This is defined as time from the date of randomization to the first day of a platelet transfusion-free period lasting at least 8 weeks.
Duration of platelet transfusion independence | Year 1, Year 2
  This is defined for participants who have achieved platelet transfusion independence only and will be calculated from the first date of platelet transfusion-free resulting in achievement of transfusion independence to the date before becoming platelet transfusion dependent.
Percentage of participants with platelet transfusion independence | Year 1, Year 2
  Platelet transfusion independence is defined as the absence of platelet transfusion for at least 8 weeks. Platelet count should be higher than the baseline count.
Percentage of participants with platelet transfusion frequency reduction at Week 24 | Week 24
  This is defined as a reduction by at least 50 percent during the 4 prior weeks as compared to the 4 weeks prior to randomization.
Percentage of participants with platelet response (Hematologic improvement (HI) - platelet)) | Week 24, Year 1, Year 2
  Platelet response is defined as HI-platelet per International Working Group criteria.
Time to platelet response | Week 24, Year 1, Year 2
  This is defined as time from the date of randomization to the first date of achieving the platelet response criteria per modified IWG criteria.
Duration of platelet response | Week 24, Year 1, Year 2
  This is defined for participants who have achieved platelet response and will be calculated from the first date of achieving the platelet response criteria to the date before loss of platelet response per modified IWG criteria.
Percentage of hematologic improvement-erythroid and -neutrophil | Week 24, Year 1, Year 2
  per modified IWG criteria at 24 weeks, Year 1 and 2
Percentage of participants with disease progression excluding relapse after HI | Week 24, Year 1, Year 2
  This is with regards to blast counts for both investigator assessment and central review per modified IWG criteria.
Percentage of participants with relapse after HI and transfusion independence | Week 24, Year 1, Year 2
  The percentage of participants with relapse after HI and transfusion independence at Week 24, Year 1 and 2.
Percentage of participants with progression to Acute myeloid leukemia (AML) | Week 24, Year 1, Year 2
  This is defined as ≥ 20% blasts at Week 24, Year 1 and 2 for both investigator assessment and central review per WHO classification revised 4th edition.
Leukemia free survival (LFS) | Week 24, Year 1, Year 2
  This is defined as time from the date of randomization to progression to AML per WHO classification revised 4th edition of ≥ 20 percent blasts or death due to any cause for both investigator assessment and central review.
Clinically significant bleeding events | Week 24, Year 1, Year 2
  This is defined as ≥ grade 2 events as per WHO bleeding scale.
Overall survival (OS) | Week 24, Year 1, Year 2
  OS is defined as time from randomization to death due to any cause.
Quality of Life measured using QLQ-C30 | Baseline, every 4 weeks until week 52, every 8 weeks after week 52 up to end of treatment or end of post-treatment follow-up, approximately 3.5 years.
  The changes from baseline to each visit where measured using QLQ-C30. EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Subject's responses to 28 questions about their physical functioning, disease symptoms, global health status and utilities are scored on a 4-point scale (1=Not at all to 4=Very much), a low score indicates a high / healthy level of functioning. And the responses to 2 questions about health-related QoL are scored on a 7-point scale (1=Very poor to 7=Excellent), a high score indicates a high / healthy level of functioning.
  Using linear transformation, raw scores are standardized, so that scores range from 0 to 100.
Pharmacokinetics (PK): Cmax | Intensive: pre-dose, 1, 2, 4, 6, 8, and 24 hours post-dose. Trough: 15th days after starting the initial dose or each dose modification until reaching the maximum dose.
  Full PK profile of eltrombopag over 24 hours at steady state at the initial dose, and at 125 mg and 150 mg when applicable, in subset of participants.
PK: Tmax | Intensive: pre-dose, 1, 2, 4, 6, 8, and 24 hours post-dose. Trough: 15th days after starting the initial dose or each dose modification until reaching the maximum dose.
  Full PK profile of eltrombopag over 24 hours at steady state at the initial dose, and at 125 mg and 150 mg when applicable, in subset of participants.
PK: AUC | Intensive: pre-dose, 1, 2, 4, 6, 8, and 24 hours post-dose. Trough: 15th days after starting the initial dose or each dose modification until reaching the maximum dose.
  Full PK profile of eltrombopag over 24 hours at steady state at the initial dose, and at 125 mg and 150 mg when applicable, in subset of participants.
Trough concentrations of eltrombopag at steady state | Intensive: pre-dose, 1, 2, 4, 6, 8, and 24 hours post-dose. Trough: 15th days after starting the initial dose or each dose modification until reaching the maximum dose.
  at each dose level in all the participants

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- Japan (20):
  - Novartis Investigative Site, Narita, Chiba
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Ohtake, Hiroshima
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Itabashi Ku, Tokyo
  - Novartis Investigative Site, Shimonoseki, Yamaguchi
  - Novartis Investigative Site, Aomori
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Gifu
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com